CLINICAL TRIAL: NCT00379145
Title: A Phase II Evaluation of Trabectedin (Yondelis, R279741) in the Treatment of Advanced, Persistent, or Recurrent Uterine Leiomyosarcomas
Brief Title: Trabectedin in Treating Patients With Advanced, Persistent, or Recurrent Leiomyosarcoma of the Uterus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0087M; CDR0000502192 (Other: CDR); NCI-2009-00573 (Other: NCI)
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2015-05

CONDITIONS: Sarcoma
Keywords: uterine leiomyosarcoma; recurrent uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trabectedin (Experimental): Trabectedin IV over 24 hours every 3 weeks
  Interventions: Drug: trabectedin

INTERVENTIONS:
Drug: trabectedin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as trabectedin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well trabectedin works in treating patients with advanced, persistent, or recurrent leiomyosarcoma of the uterus.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of trabectedin, as measured by frequency and duration of objective response, in patients with advanced, persistent, or recurrent uterine leiomyosarcoma.
* Determine the nature and degree of toxicity of this drug in these patients.

OUTLINE: This is a nonrandomized, multicenter study.

Patients receive trabectedin IV continuously over 24 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients who achieve a confirmed complete response may receive at least 2 additional courses.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 43 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed uterine leiomyosarcoma

  * Histological confirmation of original primary tumor required
* Advanced, persistent, or recurrent disease

  * Documented disease progression
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques, including palpation, plain x-ray, CT scan, and MRI OR ≥ 10 mm by spiral CT scan

  * At least 1 target lesion

    * Tumors within a previously irradiated field are considered nontarget lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiotherapy
* Ineligible for a higher priority GOG protocol (i.e., any active phase III GOG protocol for the same patient population)

PATIENT CHARACTERISTICS:

* GOG performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Platelet count ≥ 100,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Hemoglobin > 9.0 g/dL
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin normal
* AST ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 1.5 times ULN
* CPK ≤ ULN
* No active infection requiring antibiotics (except for patients with uncomplicated UTI)
* No neuropathy (sensory or motor) > grade 1
* No other invasive malignancy within the past 5 years except for nonmelanoma skin cancer
* No known active liver disease or hepatitis
* Must be willing/able to have a central venous catheter

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior surgery, radiotherapy, or other therapy
* No prior cancer treatment that would preclude study therapy
* No prior cytotoxic chemotherapy or biologic therapy for uterine sarcoma
* No prior chemotherapy for any abdominal or pelvic tumor within the past 5 years

  * Prior adjuvant chemotherapy for localized breast cancer is allowed provided it was completed more than 3 years ago and there is no evidence of recurrent or metastatic disease
* No prior trabectedin
* No prior radiotherapy within the past 5 years to any portion of the abdominal cavity or pelvis other than for treatment of uterine sarcoma

  * Prior radiotherapy for localized cancer of the breast, head and neck or skin is allowed, provided that it was completed more than 3 years ago and there is no evidence of recurrent or metastatic disease
* At least 1 week since prior hormonal therapy for the malignancy (continuation of hormone replacement therapy is permitted)
* No concurrent amifostine or other protective agents

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-06; Primary Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley J. Monk, MD, Study Chair — Chao Family Comprehensive Cancer Center
Locations (32):
- United States (32):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - St. John's Regional Health Center, Springfield, Missouri
  - Women's Cancer Center - Lake Mead, Las Vegas, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Background] Tewari D, Saffari B, Cowan C, Wallick AC, Koontz MZ, Monk BJ. Activity of trabectedin (ET-743, Yondelis) in metastatic uterine leiomyosarcoma. Gynecol Oncol. 2006 Sep;102(3):421-4. doi: 10.1016/j.ygyno.2006.04.025. Epub 2006 Jun 23. PMID 16797679
- [Result] Monk BJ, Blessing JA, Street DG, Muller CY, Burke JJ, Hensley ML. A phase II evaluation of trabectedin in the treatment of advanced, persistent, or recurrent uterine leiomyosarcoma: a gynecologic oncology group study. Gynecol Oncol. 2012 Jan;124(1):48-52. doi: 10.1016/j.ygyno.2011.09.019. Epub 2011 Oct 13. PMID 21996263

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was opened to patient entry on June 4, 2007 and was closed to accrual on November 3, 2008.
Groups:
- Trabectidin: Trabectedin 1.5 mg/m2 IV over 24 hours every 3 weeks (one cycle) until disease progression or adverse effects prohibit further therapy
Period: Overall Study
Arm/Group | Trabectidin
Started | 20
Completed (Eligible and treated patients) | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Trabectidin
Number analyzed (Participants) | 20
Age, Customized [Count of Participants; unit: Participants]
  <40 years | 1
  40-49 years | 3
  50-59 years | 5
  60-69 years | 7
  70-79 years | 3
  >79 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Objective Tumor Response Rate (Complete Response [CR] or Partial Response [PR]) Using RECIST Version 1.0
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: CT scan or MRI if used to follow lesion for measurable disease every other cycle until disease progression for up to 5 years.
Population: Eligible and treated patients
Measure: Number; unit: participants
Arm/Group | Trabectidin
Number analyzed (Participants) | 20
participants
  Partial response | 2
  Complete response | 0

2. Primary Outcome: Incidence of Adverse Effects as Assessed by Common Terminology Criteria for Adverse Events Version 3.0
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up
Population: Eligible and treated patients
Measure: Number; unit: participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 3.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
- Grade 2 (CTCAE v 3.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
- Grade 3 (CTCAE v 3.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
- Grade 4 (CTCAE v 3.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
Arm/Group | Grade 0 | Grade 1 (CTCAE v 3.0) | Grade 2 (CTCAE v 3.0) | Grade 3 (CTCAE v 3.0) | Grade 4 (CTCAE v 3.0)
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
participants
  Leukopenia | 2 | 0 | 7 | 10 | 1
  Thrombocytopenia | 13 | 4 | 0 | 3 | 0
  Neutropenia | 2 | 0 | 2 | 11 | 5
  Anemia | 3 | 10 | 6 | 1 | 0
  Other hematologic | 18 | 0 | 2 | 0 | 0
  Coagulation | 19 | 1 | 0 | 0 | 0
  Hemorrhage | 18 | 2 | 0 | 0 | 0
  Nausea | 3 | 11 | 6 | 0 | 0
  Vomiting | 7 | 10 | 3 | 0 | 0
  Bilirubin | 19 | 1 | 0 | 0 | 0
  ALT | 9 | 4 | 5 | 2 | 0
  Alkaline Phosphatase | 19 | 1 | 0 | 0 | 0
  Dermatologic | 14 | 4 | 2 | 0 | 0
  Infection | 17 | 0 | 2 | 1 | 0
  Pulmonary | 15 | 4 | 1 | 0 | 0
  Metabolic | 8 | 5 | 4 | 3 | 0
  Lymphatics | 16 | 4 | 0 | 0 | 0
  Pain | 8 | 10 | 2 | 0 | 0
  Constitutional | 17 | 3 | 0 | 0 | 0
  Fatigue | 5 | 8 | 7 | 0 | 0
  Musculoskeletal | 15 | 4 | 1 | 0 | 0
  Neurotoxicity | 16 | 4 | 0 | 0 | 0
  Peripheral neuropathy | 18 | 2 | 0 | 0 | 0
  Renal | 19 | 1 | 0 | 0 | 0
  Ocular | 16 | 3 | 1 | 0 | 0
  Vascular | 19 | 0 | 0 | 1 | 0
  Flu-like syndrome | 19 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up
Arm/Group | Trabectidin
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectidin (N=20)
Neutrophils (Blood and lymphatic system disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Neck Nos (Infections and infestations) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectidin (N=20)
Rhinitis (Immune system disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Neutrophils (Blood and lymphatic system disorders) | 18
Platelets (Blood and lymphatic system disorders) | 8
Leukocytes (Blood and lymphatic system disorders) | 18
Lymphopenia (Blood and lymphatic system disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 17
Palpitations (Cardiac disorders) | 1
Cardiac Arrhythmia - Other (Cardiac disorders) | 1
Ventricular Arrhythmia - Tachycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 1
Cardiac General - Other (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 1
Inr (Vascular disorders) | 2
Ptt (Vascular disorders) | 1
Weight Gain (General disorders) | 4
Fever (General disorders) | 2
Weight Loss (General disorders) | 2
Rigors/Chills (General disorders) | 1
Fatigue (General disorders) | 16
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1
Bruising (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Flushing (Skin and subcutaneous tissue disorders) | 2
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Hot Flashes (Endocrine disorders) | 3
Flatulence (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Distention (Gastrointestinal disorders) | 1
Taste Alteration (Gastrointestinal disorders) | 2
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 13
Anorexia (Gastrointestinal disorders) | 6
Dehydration (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 17
Gastrointestinal - Other (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 8
Hemorrhage, Gi - Rectum (Vascular disorders) | 1
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 2
Febrile Neutropenia (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Pharynx (Infections and infestations) | 1
Edema: Limb (Blood and lymphatic system disorders) | 5
Edema: Head And Neck (Blood and lymphatic system disorders) | 1
Ast (Metabolism and nutrition disorders) | 10
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 3
Cholesterol,serum High (Metabolism and nutrition disorders) | 1
Proteinuria (Metabolism and nutrition disorders) | 2
Creatinine (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Alt (Metabolism and nutrition disorders) | 12
Alkaline Phosphatase (Metabolism and nutrition disorders) | 1
Bilirubin (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Cpk (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 2
Muscle Weakness - Extremity-Upper (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 3
Neurology - Other (Nervous system disorders) | 2
Mood Alteration - Depression (Nervous system disorders) | 4
Mood Alteration - Anxiety (Nervous system disorders) | 2
Mood Alteration - Agitation (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Neuropathy-Sensory (Nervous system disorders) | 5
Neuropathy-Motor (Nervous system disorders) | 2
Ocular/Visual - Other (Eye disorders) | 1
Flashing Lights/Floaters (Eye disorders) | 1
Blurred Vision (Eye disorders) | 3
Pain - Other (General disorders) | 1
Pain: Pelvis (General disorders) | 2
Pain: Chest /Thorax Nos (General disorders) | 1
Pain: Chest Wall (General disorders) | 2
Pain: Throat/Pharynx/Larynx (General disorders) | 2
Pain: Head/Headache (General disorders) | 9
Pain: Neck (General disorders) | 2
Pain: Extremity-Limb (General disorders) | 6
Pain: Back (General disorders) | 3
Pain: Joint (General disorders) | 5
Pain: Stomach (General disorders) | 1
Pain: Oral Cavity (General disorders) | 3
Pain: Abdominal Pain Nos (General disorders) | 3
Pain: Liver (General disorders) | 1
Pain: Muscle (General disorders) | 3
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Renal/Genitourinary - Other (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1
Flu-Like Syndrome (General disorders) | 1
Vascular - Other (Vascular disorders) | 1
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 2
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less